CLINICAL TRIAL: NCT03437746
Title: Impact of Preoperative Single Corticosteroid Flash on Morbidity After Colorectal Resection: Monocentric Prospective Pilot Study
Acronym: CORTICOLON
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient rate of inclusion
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOUSSOT AOI 2017
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Elective Colorectal Surgery
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: injection of methylprednisolone at anesthetic induction — intravenous administration : 20 mg/kg, over 30 minutes at anesthetic induction
Biological: Blood samples — Blood samples (D0, D1, D2, D3, D4)

SUMMARY:
Complications due to infection after colorectal surgery are frequent, affecting up to 25% of patients. Infection increases mortality, lengthens hospital stays, increases costs and decreases long term survival for cancer patients. Perioperative inflammation leads to hypercatabolism, denutrition and immunosuppression, all of which are associated to postoperative infection. Data from various sources suggests that modulating perioperative inflammatory response through the injection of corticosteroids would benefit the patient by reducing the number of postoperative complications after major surgery. Pre- or perioperative intravenous administration of a single corticosteroid flash is a means of modulating systemic inflammation that has been suggested for numerous types of surgeries, including pancreatic surgery. The objective of this study is to assess whether a preoperative single corticosteroid flash (methylprednisolone: 20 mg/kg IV at anesthetic induction) reduces the risk of serious complications after elective colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient undergoing elective colorectal surgery (diverticulitis, malignant or benign tumor, inflammatory intestinal disease, re-establishing continuity, endometriosis, or other)
* Bowel continuity is restored immediately after surgery, with or without a protective stoma.
* Patient with proper understanding who has been informed about the study, and who has consented to being part of the study

Exclusion Criteria:

* Adult under guardianship
* Patient who is not covered under the national health system
* Women who are pregnant or breastfeeding
* Colorectal resection with concomitant hyperthermic intraperitoneal chemotherapy
* Patient under long term corticosteroid therapy
* Preoperative natremia > 147 mmol/L
* Hypokalemia (< 3,3 mmol/L)
* Patient with a contraindication to Methylprednisolone Mylan® :

  * Active infection
  * Active viral disease (namely hepatitis, herpes, varicella, shingles),
  * A psychotic condition that is not currently treated with medication,
  * Vaccination with a live vaccine or live attenuated within the last 3 months,
  * Hypersensitivity to methylprednisolone or to any of the excipients found in Methylprednisolone Mylan®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Frequency of postoperative complications, occuring up to 30 days post-operatively | Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Evaluation of pre-operative high dose corticosteroids in elective colorectal surgery and effects on gut barrier function : A phase 2 clinical trial